CLINICAL TRIAL: NCT07266831
Title: A Phase 2/3, Randomized, Active-Controlled, Open-Label (Phase 2) and Double-Blind (Phase 3) Study to Evaluate the Antiretroviral Activity, Safety, and Tolerability of Islatravir (ISL) and Ulonivirine (ULO) Once Weekly Compared With Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) Once Daily in Treatment-Naïve Adult Participants Living With HIV-1
Brief Title: A Clinical Study of Islatravir and Ulonivirine for People With HIV-1 Who Have Not Been Treated Before (MK-8591B-062)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591B-062; U1111-1323-4689 (Registry Identifier: UTN); 2025-522519-40 (Registry Identifier: EU CT); MK-8591B-062 (Other: MSD)
Record Dates: First submitted 2025-12-01; First posted 2025-12-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — islatravir; ulonivirine; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2: no masking Phase 3: Participant, Sponsor, and Investigator are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2: ISL + ULO (Experimental): Islatravir (ISL) 2mg and Ulonivirine (ULO) 200mg administered orally once weekly (qw) for 96 weeks
  Interventions: Drug: ISL; Drug: ULO
- Phase 2: BIC/FTC/TAF (Active Comparator): Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) 50/200/25 mg, administered orally once daily (qd) for 96 weeks
  Interventions: Drug: BIC/FTC/TAF
- Phase 3: ISL/ULO and Placebo to BIC/FTC/TAF (Experimental): ISL/ULO fixed dose combination (2/200 mg), administered orally qw, and matching placebo to BIC/FTC/TAF administered orally qd for 96 weeks
  Interventions: Drug: Placebo for BIC/FTC/TAF; Drug: ISL/ULO
- Phase 3: BIC/FTC/TAF and Placebo to ISL/ULO (Active Comparator): BIC/FTC/TAF 50/200/25 mg, administered orally qd, and matching placebo to ISL/ULO administered orally qw for 96 weeks
  Interventions: Drug: BIC/FTC/TAF; Drug: Placebo to ISL/ULO

INTERVENTIONS:
Drug: ISL — ISL 2 x 1 mg oral capsules administered qw for 96 weeks
  Other Names: islatravir; MK-8591
  Arms: Phase 2: ISL + ULO
Drug: ULO — ULO 2 x 100 mg oral tablets administered qw for 96 weeks
  Other Names: ulonivirine; MK-8507
  Arms: Phase 2: ISL + ULO
Drug: BIC/FTC/TAF — BIC/FTC/TAF 50/200/25 mg oral tablet administered qd for 96 weeks
  Other Names: bictegravir/emtricitabine/tenofovir alafenamide; BIKTARVY®
  Arms: Phase 2: BIC/FTC/TAF; Phase 3: BIC/FTC/TAF and Placebo to ISL/ULO
Drug: Placebo for BIC/FTC/TAF — BIC/FTC/TAF-matching placebo oral tablet administered qd for 96 weeks
  Arms: Phase 3: ISL/ULO and Placebo to BIC/FTC/TAF
Drug: Placebo to ISL/ULO — ISL/ULO-matching placebo oral tablets administered qw for 96 weeks
  Arms: Phase 3: BIC/FTC/TAF and Placebo to ISL/ULO
Drug: ISL/ULO — ISL/ULO fixed-dose combination 2 mg/200 mg oral tablet administered qw for 96 weeks
  Other Names: MK-8591B
  Arms: Phase 3: ISL/ULO and Placebo to BIC/FTC/TAF

SUMMARY:
Researchers are looking for new ways to treat HIV-1 (Human Immunodeficiency Virus Type 1). The usual (standard) treatment for HIV-1 is antiretroviral therapy (ART), which includes taking medicines to lower the amount of HIV-1 in the body. Standard ART helps people live longer, but people must take up to 3 medicines up to twice a day. Standard ART may also cause other health problems. Researchers want to know if a study ART works as well as a standard ART to treat HIV-1. The study ART combines 2 medicines, islatravir and ulonivirine, and is taken once a week. The goals of this study are to learn: 1) If the study ART works as well as a standard ART to treat HIV-1, and 2) About the safety of the study ART and if people tolerate it compared to a standard ART.

ELIGIBILITY:
Inclusion Criteria:

* Phase 2: Is human immunodeficiency virus type 1 (HIV-1) positive with Plasma HIV-1 ribonucleic acid (RNA) ≥500 and ≤100,000 copies/mL.
* Phase 3: Is HIV-1 positive with Plasma HIV-1 RNA ≥500 copies/mL.
* Phase 2: Has cluster of differentiation 4-positive (CD4+) T-cell count ≥200 cells/mm^3.
* Is naïve to antiretroviral therapy (ART), defined as having received no prior therapy with any antiretroviral agent following a diagnosis of HIV 1 infection.

Exclusion Criteria:

* Has human immunodeficiency virus type 2 (HIV-2) infection.
* Has a diagnosis of an active acquired immune deficiency syndrome (AIDS)-defining opportunistic infection.
* Has active hepatitis C virus (HCV) or active hepatitis B virus (HBV) infection.
* Has a history of malignancy ≤5 years prior to providing documented informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or in situ anal cancer, or cutaneous Kaposi's sarcoma.
* Has prior exposure to islatravir (ISL) or ulonivirine (ULO) for any duration any time prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2029-10-05 (Estimated); Study Completion 2030-04-25 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Percentage of Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/mL at Week 24 | Week 24
  Plasma HIV-1 ribonucleic acid (RNA) quantification will be performed at the central laboratory using a polymerase chain reaction (PCR) assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 24.
Phase 2: Percentage of Participants Who Experience an Adverse Event (AE) at Week 24 | Week 24
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 2: Percentage of Participants Who Discontinue Study Intervention Due to an AE at Week 24 | Week 24
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 3: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 48.
Phase 3: Percentage of Participants Who Experience an AE at Week 48 | Week 48
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 3: Percentage of Participants Who Discontinue Study Intervention Due to an AE at Week 48 | Week 48
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

SECONDARY OUTCOMES:
Phase 2: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 48.
Phase 2: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 96.
Phase 2: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 24 | Week 24
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 24.
Phase 2: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 48.
Phase 2: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 96.
Phase 2: Mean Change From Baseline in Cluster of Differentiation 4-Positive (CD4+) T-Cell Count at Week 24 | Baseline (Day 1) and Week 24
  Blood samples will be collected to measure CD4+ T-cell count. The mean change from baseline in CD4+ T-cell count will be calculated at 24 weeks.
Phase 2: Mean Change From Baseline in CD4+ T-Cell Count at Week 48 | Baseline (Day 1) and Week 48
  Blood samples will be collected to measure CD4+ T-cell count. The mean change from baseline in CD4+ T-cell count will be calculated at 48 weeks.
Phase 2: Mean Change From Baseline in CD4+ T-Cell Count at Week 96 | Baseline (Day 1) and Week 96
  Blood samples will be collected to measure CD4+ T-cell count. The mean change from baseline in CD4+ T-cell count will be calculated at 96 weeks.
Phase 2: Percentage of Participants Who Experience an AE | Up to approximately 102 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 2: Percentage of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 96 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 2: Number of Participants With Evidence of Viral Drug Resistance-Associated Substitutions at Week 24 | Week 24
  Participants who meet the definition of clinically significant confirmed viremia (CSCV) or who discontinue study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation, will be assessed for development of viral drug resistance. Among such participants, those with confirmed HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses set. In addition, anyone for whom available genotypic and/or phenotypic data show evidence of resistance, irrespective of viral load, will also be included in the resistance analyses set. The number of participants in each treatment group who have evidence of resistance-associated substitutions at week 24 will be presented.
Phase 2: Number of Participants With Evidence of Viral Drug Resistance-Associated Substitutions at Week 48 | Week 48
  Participants who meet the definition of clinically significant confirmed viremia (CSCV) or who discontinue study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation, will be assessed for development of viral drug resistance. Among such participants, those with confirmed HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses set. In addition, anyone for whom available genotypic and/or phenotypic data show evidence of resistance, irrespective of viral load, will also be included in the resistance analyses set. The number of participants in each treatment group who have evidence of resistance-associated substitutions at week 48 will be presented.
Phase 2: Number of Participants With Evidence of Viral Drug Resistance-Associated Substitutions at Week 96 | Week 96
  Participants who meet the definition of clinically significant confirmed viremia (CSCV) or who discontinue study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation, will be assessed for development of viral drug resistance. Among such participants, those with confirmed HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses set. In addition, anyone for whom available genotypic and/or phenotypic data show evidence of resistance, irrespective of viral load, will also be included in the resistance analyses set. The number of participants in each treatment group who have evidence of resistance-associated substitutions at week 96 will be presented.
Phase 3: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 96.
Phase 3: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 48.
Phase 3: Percentage of Participants With HIV-1 RNA <200 Copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 96.
Phase 3: Mean Change From Baseline in Cluster of Differentiation 4-Positive (CD4+) T-Cell Count at Week 48 | Baseline (Day 1) and Week 48
  Blood samples will be collected to measure CD4+ T-cell count. The mean change from baseline in CD4+ T-cell count will be calculated at 48 weeks.
Phase 3: Mean Change From Baseline in Cluster of Differentiation 4-Positive (CD4+) T-Cell Count at Week 96 | Baseline (Day 1) and Week 96
  Blood samples will be collected to measure CD4+ T-cell count. The mean change from baseline in CD4+ T-cell count will be calculated at 96 weeks.
Phase 3: Percentage of Participants Who Experience an AE | Up to approximately 102 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 3: Percentage of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 96 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Phase 3: Number of Participants With Evidence of Viral Drug Resistance-Associated Substitutions at Week 48 | Week 48
  Participants who meet the definition of clinically significant confirmed viremia (CSCV) or who discontinue study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation, will be assessed for development of viral drug resistance. Among such participants, those with confirmed HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses set. In addition, anyone for whom available genotypic and/or phenotypic data show evidence of resistance, irrespective of viral load, will also be included in the resistance analyses set. The number of participants in each treatment group who have evidence of resistance-associated substitutions at week 48 will be presented.
Phase 3: Number of Participants With Evidence of Viral Drug Resistance-Associated Substitutions at Week 96 | Week 96
  Participants who meet the definition of clinically significant confirmed viremia (CSCV) or who discontinue study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation, will be assessed for development of viral drug resistance. Among such participants, those with confirmed HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses set. In addition, anyone for whom available genotypic and/or phenotypic data show evidence of resistance, irrespective of viral load, will also be included in the resistance analyses set. The number of participants in each treatment group who have evidence of resistance-associated substitutions at week 96 will be presented.
Phase 3: Mean Change From Baseline in Body Weight at Week 48 | Baseline (Day 1) and Week 48
  Body weight will be collected throughout the study.
Phase 3: Mean Change From Baseline in Body Weight at Week 96 | Baseline (Day 1) and Week 96
  Body weight will be collected throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (21):
- United States (18):
  - Vivent Health ( Site 1519), Denver, Colorado
  - Whitman-Walker Institute ( Site 1538), Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 1503), Ft. Pierce, Florida
  - CAN Community Health- Miami Gardens ( Site 1549), Miami, Florida
  - Orlando Immunology Center ( Site 1501), Orlando, Florida
  - CAN Community Health ( Site 1510), Sarasota, Florida
  - Triple O Research Institute ( Site 1505), West Palm Beach, Florida
  - Metro Infectious Diseases Consultants L.L.C. ( Site 1509), Decatur, Georgia
  - Mercer university, Department of internal medicine-Clinical Research ( Site 1512), Macon, Georgia
  - KC CARE Health Center ( Site 1506), Kansas City, Missouri
  - ID Care ( Site 1507), Hillsborough, New Jersey
  - Regional Center for Infectious Diseases ( Site 1516), Greensboro, North Carolina
  - The Ohio State University ( Site 1536), Columbus, Ohio
  - University of Pennsylvania Perelman School of Medicine ( Site 1508), Philadelphia, Pennsylvania
  - Saint Hope Foundation, Inc. ( Site 1504), Bellaire, Texas
  - Prism Health North Texas, Oak Cliff Health Center ( Site 1514), Dallas, Texas
  - Texas Center for Infectious Disease Associates ( Site 1502), Fort Worth, Texas
  - DCOL Center for Clinical Research ( Site 1511), Longview, Texas
- Spectrum Health ( Site 3307), Vancouver, British Columbia, Canada
- Guatemala (2):
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 3801), Guatemala City
  - MEDI-K ( Site 3803), Guatemala City

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com